CLINICAL TRIAL: NCT06551324
Title: A PHASE 3, RANDOMIZED, OPEN-LABEL STUDY OF PF-06821497 (MEVROMETOSTAT) IN COMBINATION WITH ENZALUTAMIDE COMPARED WITH ENZALUTAMIDE OR DOCETAXEL IN PARTICIPANTS WITH METASTATIC CASTRATION RESISTANT PROSTATE CANCER PREVIOUSLY TREATED WITH ABIRATERONE ACETATE (MEVPRO-1)
Brief Title: A Study to Learn About the Investigational Medicine Called PF-06821497 (Mevrometostat) in Men With mCRPC Who Were Previously Treated With Abiraterone Acetate for Prostate Cancer (MEVPRO-1).
Acronym: MEVPRO-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2321014; 2024-511650-50-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-07-25; First posted 2024-08-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Keywords: Prostate cancer; Enhancer of zeste homolog 2; castrate resistant prostate cancer; Hormone resistant; Metastatic hormone resistant prostate cancer; Metastatic castrate resistant prostate cancer; PF-06821497; Enzalutamide; Docetaxel; Advanced prostate cancer; Efficacy; Safety; Open-label; Relapsed; refractory
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence | interventions — PF06821497; Docetaxel; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Investigational Arm A: PF-06821497 875 mg twice daily (BID) + enzalutamide 160 mg every day (QD)
  Interventions: Drug: PF-06821497; Drug: Enzalutamide
- Arm B (Active Comparator): Comparator Arm B: Physician's choice of enzalutamide 160 mg QD or docetaxel 75 mg/m2 intravenous (IV) every 21 days
  Interventions: Drug: Docetaxel; Drug: Enzalutamide

INTERVENTIONS:
Drug: PF-06821497 — 875 mg BID (2 times a day)
  Other Names: Mevrometostat
  Arms: Arm A
Drug: Docetaxel — 75 mg/m2 IV (every 21 days)
  Other Names: Taxotere
  Arms: Arm B
Drug: Enzalutamide — 160 mg QD
  Other Names: XTANDI

SUMMARY:
Pfizer MEVPRO-1 (C2321014) is a randomized, open-label, multi-center clinical trial evaluating whether combining the study medicine (PF-06821497) with enzalutamide is safe and effective compared to physician's choice of either second-line androgen receptor (AR) directed therapy with enzalutamide or docetaxel (chemotherapy) for treating metastatic castration-resistant prostate cancer (mCRPC) after progression on prior abiraterone acetate treatment.

The primary objective of this clinical trial is to assess the radiographic progression free survival (rPFS) of the combination of PF-06821497 plus enzalutamide versus physician's choice of enzalutamide or docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features.
* Metastatic disease in bone documented on bone scan, or in soft tissue documented on CT/MRI scan.
* Progressive disease in the setting of surgical or medical castration with evidence of disease progression on treatment with abiraterone acetate in the mCSPC setting or first line mCRPC setting is required.
* Eastern Cooperate Oncology Group (ECOG) performance status 0 - 2, with life expectancy of at least 6 months as assessed by the investigator.

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may make the participant inappropriate for the study.
* Know history of active inflammatory gastrointestinal disease, chronic diarrhea, or previous gastric resection or lap-band surgery.
* Clinically significant cardiovascular disease.
* Known or suspected brain metastasis or active leptomeningeal disease or clinically significant history of seizure.
* Prior treatment for prostate cancer at any stage with any cytotoxic chemotherapy, radioligand therapy (i.e. 177Lu-PSMA-617, radium 223), androgen receptor signaling inhibitors (ARSi) including enzalutamide, apalutamide, darolutamide, poly ADP-ribose polymerase (PARP) monotherapy or other systemic anti-cancer treatment, with the following exceptions:

  1. Treatment with first-generation antiandrogen agents, if discontinued prior to first dose of study intervention.
  2. Docetaxel treatment is allowed for mCSPC, as long as no signs of failure, or disease progression occurred during treatment or within 3 months of treatment completion.
* Previous administration with an investigational product within 30 days or 5 half-lives preceding the first dose of study intervention (whichever is shorter).
* Inadequate organ function.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2028-10-29 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) assessed by blinded independent central review (BICR) per RECIST v1.1 and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) | Randomization up to approximately 2 years.
  rPFS is defined as the time from the date of randomization to first objective evidence of radiographic progression as assessed in soft tissue per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or in bone per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines by BICR, or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Randomization up to approximately 4.5 years.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Objective Response (ORR) | Randomization up to approximately 2 years.
  The objective response rate is defined as the proportion of participants with measurable soft tissue disease at baseline who have a confirmed objective response of complete response (CR) or partial response (PR) per RECIST v1.1.
Duration of Response (DoR) in measurable soft tissue disease | Randomization up to approximately 2 years.
  The DoR is defined as the first objective evidence of soft tissue response (CR or PR, whichever is earlier) to radiographic progression or death due to any cause whichever occurs first.
Time to prostate specific antigen (PSA) progression. | Randomization up to approximately 2 years.
  Proportion of participants with PSA response ≥50% in participants with detectable PSA values at baseline.
Time to initiation of antineoplastic therapy. | Randomization up to approximately 4.5 years.
  Time from randomization to first use of new antineoplastic therapy.
Prostate Specific Antigen Response | Randomization up to approximately 2 years.
  Proportion of participants with PSA response ≥50% in participants with detectable PSA values at baseline.
Incidence of Adverse Events | Randomization up to approximately 4.5 years
  Type, incidence, severity [as graded by National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) v5.0], seriousness and relationship to study medications of AEs.
Time to first symptomatic skeletal event | Randomization up to approximately 2 years.
  Time from randomization to first symptomatic skeletal event (symptomatic bone fractures, spinal cord compression, surgery or radiation to the bone whichever is first).
Change from baseline in patient reported pain symptoms per Brief Pain Inventory-Short Form (BPI-SF) | Randomization up to approximately 4.5 years
  Analysis of Brief Pain Inventory-Short Form (BPI-SF) will be based on the pain severity score (mean of individual BPI-SF items 3, 4, 5 and 6), the pain interference score (mean of items 9A-9G), and the single BPI-SF Item 3 which asks the patient to rate pain at its worst in the last 24 hours.
Change from baseline in health-related quality of life (HRQoL) per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization to approximately 4.5 years
  Change from baseline in HRQoL (FACT-P total score) will be presented. The FACT-P total score will be calculated based on the participant responses to the 39 items in the FACT-P questionnaire. Each item is rated on a 0 to 4 Likert-type scale and then combined to produce the FACT-P total score (0-156), with higher scores representing better health-related quality of life.
Change from baseline in social/family well-being per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization up to approximately 4.5 years
  Change from baseline in social/family well-being score will be presented. The social/family well-being score will be calculated based on 7 items in the FACT-P questionnaire; score range 0-28. Each item is rated on a 0 to 4 Likert-type scale
Change from baseline in emotional well-being per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization up to approximately 4.5 years
  Change from baseline in emotional well-being score will be presented. The emotional well-being score will be calculated based on 6 items in the FACT-P questionnaire; score range 0-24. Each item is rated on a 0 to 4 Likert-type scale
Change from baseline in functioning well-being per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization up to approximately 4.5 years
  Change from baseline in functioning well-being score will be presented. The functioning well-being score will be calculated based on 7 items in the FACT-P questionnaire; score range 0-28. Each item is rated on a 0 to 4 Likert-type scale
Change from baseline in physical well-being per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization to approximately 4.5 years
  Change from baseline in physical well-being score will be presented. The physical well-being score will be calculated based on 7 items in the FACT-P questionnaire; score range 0-28. Each item is rated on a 0 to 4 Likert-type scale
Change from baseline in symptoms per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization up to approximately 4.5 years
  Change from baseline prostate cancer symptoms (PCS) score will be presented. The PCS score will be calculated based on 12 items in the FACT-P questionnaire; score range 0-48. Each item is rated on a 0 to 4 Likert-type scale
Change from baseline in patient reported health status per European Quality of Life 5-Dimension 5 Level (EQ-5D-5L) | Randomizaton up to approximately 4.5 years
  Participants will self-rate their current state of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression by choosing 1 of 5 possible responses that record the level of severity (no problems, slight problems, moderate problems, severe problems, or extreme problems) within each dimension. The questionnaire also includes a visual analog scale to self-rate general health state on a scale from "the worst health you can imagine" to "the best health you can imagine."
Symptomatic toxicity as measured by items from the Patient-Reported Outcome CTCAE (PRO-CTCAE) | Randomization up to approximately 4.5 years
  Each selected PRO-CTCAE items will be assessed related to one or more attributes that include counts for the frequency, severity, and/or interference with usual or daily activities.
Overall side effect burden as measured by the FACT- GP5 | Randomization to approximately 4.5 years
  The FACT-GP5 question assesses overall side effect burden with the following response options "I am bothered by side effects of treatment," is rated on a 5-point scale ranging from "not at all" (0) to "very much" (4) and counts will be presented.
Time to confirmatory deterioration in patient-reported pain symptoms per BPI-SF Item 3 "worst pain in 24 hours" | Randomization up to approximately 4.5 years
  Defined as the time from randomization to onset of pain progression, which is defined as > 2-point increase from baseline in the score from the BPI-SF Question 3 that is confirmed at the next consecutive assessment > 4 weeks apart or an initial deterioration followed by death before the next assessment
Time to definitive deterioration in patient-reported health related quality of life (HRQoL) per FACT-P | Randomization up to approximately 4.5 years
  Defined as the time from randomization to onset of definitive deterioration in FACT-P total score, which is defined as >10 point decrease from baseline and no subsequent observations with a <10 point decrease from baseline FACT-P total score
Time to definitive deterioration in patient-reported physical well-being per FACT-P | Randomization up to approximately 4.5 years
  Time to definitive deterioration in physical well-being (PWB) per FACT-P is defined as the time from randomization to onset of definitive deterioration in physical well-being, which is defined as ≥3-point
To evaluate the PK of PF-06821497 when dosed with enzalutamide | Cycle 1 (each cycle is 28 days), Day 1 to last PK draw at the end of Cycle 6, Day 1.
  PK characterized by pre-dose trough and post-dose plasma concentrations of PF-06821497 at selected visits.
To assess circulating tumor DNA (ctDNA) at baseline and on treatment to evaluate tumor burden. | Baseline up to approximately 2 years.
  Evaluation of ctDNA burden at baseline and on study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (229):
- United States (66):
  - Urology Centers of Alabama, Homewood, Alabama
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - Los Angeles Cancer Network, Anaheim, California
  - UCSF Cancer Center Berkeley, Berkeley, California
  - UCSF Cancer Center Burlingame, Burlingame, California
  - Los Angeles Cancer Network, Fountain Valley, California
  - Los Angeles Cancer Network, Glendale, California
  - Los Angeles Cancer Network, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - UCSF Investigational Drug Pharmacy, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - UCSF Cancer Center San Mateo, San Mateo, California
  - Sutter Santa Rosa, Santa Rosa, California
  - Stanford Health Care Attention: Investigational Pharmacy, Stanford, California
  - Colorado Clinical Research, Lakewood, Colorado
  - University of Miami Sylvester Comprehensive Cancer Center - Aventura, Aventura, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital and Clinics - Doral, Doral, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Kendall, Kendall, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinics, UHealth Tower, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Griffin Cancer Research Building, Miami, Florida
  - Florida Cancer Specialists, N. Venice, Florida
  - Florida Cancer Specialists, Naples, Florida
  - AdventHealth Hematology and Oncology, Orlando, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Plantation, Plantation, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Duly Health and Care, Lisle, Illinois
  - NextStage Clinical Research-Chicago-(04), Lisle, Illinois
  - Duly Health and Care, Westmont, Illinois
  - The University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - New England Cancer Specialists, Topsham, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - VA St. Louis Health Care System, St Louis, Missouri
  - AtlantiCare, Egg Harbor, New Jersey
  - Circuit Clinical /Crystal Run Healthcare LLP, Middletown, New York
  - Circuit Clinical, Middletown, New York
  - Crystal Run Healthcare, Monroe, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - Salisbury VA Medical Center, Salisbury, North Carolina
  - The Centers for Advanced Urology, LLP d/b/a Keystone Urology Specialists, Lancaster, Pennsylvania
  - AUC Urologists, LLC, Myrtle Beach, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Grand Strand Medical Center, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - USA Clinical Trials, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
- Argentina (9):
  - Centro de Urología (CDU), CABA, Buenos Aires
  - Hospital Sirio Libanes, Capital Federal, Buenos Aires
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Imagenes Mdq, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - IMAXE, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC), Buenos Aires
- Australia (3):
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Brazil (9):
  - Hospital São Carlos, Fortaleza, Ceará
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
- China (26):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Lanzhou university second hospital, Lanzhou, Gansu
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People' Hospital, Xi'an, Shaanxi
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The first affiliated hospital of Ningbo university, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (6):
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Multiscan, Pardubice, Pardubický kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha 10
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Nukleární Medicína, Hradec Králové
  - Radiodiagnostika Pardubice, Pardubice
- France (15):
  - Centre Antoine Lacassagne, Nice, Alpes-maritimes
  - Centre Antoine-Lacassagne, Nice, Alpes-maritimes
  - Centre Leon Berard, Lyon Cedex08, Auvergne-Rhône-Alpes
  - Hopitaux Universitaire de Strasbourg - Hopital Hautepierre, Strasbourg, Bas-rhin
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Brittany Region
  - CHRU de Brest, Brest, Finistère
  - Centre Hospitalier Universitaire de Nîmes - Institut de Cancérologie du Gard - Hôpital Universitaire, Nîmes, GARD
  - Oncopole Claudius Regaud, Toulouse, Haute-garonne
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - Hôpital Foch, Suresnes, Hauts-de-seine
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire, Ille-et-vilaine
  - Institut Jean Godinot, Reims, Marne
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Gustave Roussy, Villejuif, Val-de-marne
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand
- Germany (5):
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Urologie Neandertal - Praxis Mettmann, Mettmann, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Greece (4):
  - Alexandra General Hospital of Athens, Athens, Attikí
  - Athens Medical Center, Athens, Attikí
  - Metropolitan General Hospital, Athens, Attikí
  - University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí
- Hungary (2):
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Országos Onkológiai Intézet, Budapest, Pest County
- Italy (3):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - Ospedale San Raffaele, Milan
- Japan (15):
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - The University of Osaka Hospital, Suita, Osaka
  - Keio university hospital, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka International Cancer Institute, Osaka
  - Yamagata University Hospital, Yamagata
- Netherlands (4):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Tergooi MC, Hilversum, North Holland
  - Frisius Medisch Centrum, Leeuwarden, Provincie Friesland
  - Meander Medisch Centrum, Amersfoort, Utrecht
- Poland (7):
  - Regionalny Szpital Specjalistyczny im. dr. Władyslawa Biegańskiego, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw, Lower Silesian Voivodeship
  - SP ZOZ Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego w Opolu, Opole, Opole Voivodeship
  - Szpital Wojewódzki im. Mikołaja Kopernika w Koszalinie, Koszalin
- Slovakia (5):
  - Narodny onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - MILAB, s.r.o., Urologicka ambulancia, Prešov
  - BEKY - MED, s.r.o., Prešov
  - Fakultna nemocnica Trnava, Trnava
- South Africa (4):
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - Wits Clinical Research, Johannesburg, Gauteng
  - Wilgers Oncology Centre, Pretoria, Gauteng
  - TASK Eden, George, Western Cape
- South Korea (8):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-kwangyǒkshi
- Spain (10):
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Södersjukhuset, Stockholm, Stockholms LÄN [se-01]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands LÄN [se-14]
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (10):
  - Koç Üniversitesi Hastanesi, Istanbul, İ̇stanbul
  - Istanbul Universitesi Cerrahpasa, Istanbul, İ̇stanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul, İ̇stanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul, İ̇stanbul
  - I.E.U. Medical Point Hastanesi, Izmir, İ̇zmir
  - Adana City Hospital, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Ankara University Health Practice and Research Hospitals, Ankara
- United Kingdom (6):
  - Royal Blackburn Hospital, Blackburn, Blackburn WITH Darwen
  - Mid and South Essex NHS Foundation Trust, Chelmsford, Essex
  - Western General Hospital, Edinburgh, Midlothian
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321014
- See also: www.mevpro1.com — https://www.pfizerclinicaltrials.com/nct06551324-prostate-cancer-trial